CLINICAL TRIAL: NCT02570568
Title: Pen Torch Transillumination: Shedding Light on Difficult Venepuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/00152
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Disorder of Vein
Keywords: Venepuncture; Transillumination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional Venepuncture (Active Comparator): Veins will be identified by a combination of visualization and palpation. Once a suitable vein is localized, a tourniquet is applied (Braun® International, USA). The area of the skin to be cannulated is disinfected with an alcohol wipe (Webcol®, Covidien®, USA). For the setting of IV cannulation, a standardized 23G IV cannula is used (Introcan Safety®, Braun®, USA). Normal saline (PosiFlush® 3ml, BD®, USA) will be used for flushing the cannula after successful cannulation. For blood taking, a syringe (Terumo®, Philippines) ranging from 2ml to 20ml and a 23G needle (Venofix®, Braun®, USA) will be used. All instruments needed for venepuncture, including 4 IV cannula or 4 needles should be by the patient's bedside prior to the start of each venepuncture.
  Interventions: Procedure: Conventional Venepuncture
- Veinlite (Experimental): Placing Veinlite onto the skin will cause the outlines of the veins to show up. Once a suitable vein is localized, a tourniquet is applied (Braun® International, USA). The area of the skin to be cannulated is disinfected with an alcohol wipe (Webcol®, Covidien®, USA). For the setting of IV cannulation, a standardized 23G IV cannula is used (Introcan Safety®, Braun®, USA). Normal saline (PosiFlush® 3ml, BD®, USA) will be used for flushing the cannula after successful cannulation. For blood taking, a syringe (Terumo®, Philippines) ranging from 2ml to 20ml and a 23G needle (Venofix®, Braun®, USA) will be used. All instruments needed for venepuncture, including 4 IV cannula or 4 needles should be by the patient's bedside prior to the start of each venepuncture.
  Interventions: Device: Veinlite
- Pen-torch Transillumination (Experimental): The tips of the pen torches are pressed onto the skin, causing the silhouette of the vein to show up. Once a suitable vein is localized, a tourniquet is applied (Braun® International, USA). The area of the skin to be cannulated is disinfected with an alcohol wipe (Webcol®, Covidien®, USA). For the setting of IV cannulation, a standardized 23G IV cannula is used (Introcan Safety®, Braun®, USA). Normal saline (PosiFlush® 3ml, BD®, USA) will be used for flushing the cannula after successful cannulation. For blood taking, a syringe (Terumo®, Philippines) ranging from 2ml to 20ml and a 23G needle (Venofix®, Braun®, USA) will be used. All instruments needed for venepuncture, including 4 IV cannula or 4 needles should be by the patient's bedside prior to the start of each venepuncture.
  Interventions: Device: Pen-torch Transillumination

INTERVENTIONS:
Device: Veinlite — Veinlite is a device that emits red light. It provides a non-invasive technique of inserting intra-venous cannula. Placing it onto the skin will cause the outlines of the veins to show up.
  Arms: Veinlite
Device: Pen-torch Transillumination — Pen-torch Transillumination is a non-invasive technique that utilizes 2 pen-torches to provide illumination.The tips of the pen torches are pressed onto the skin, causing the silhouette of the vein to show up
  Arms: Pen-torch Transillumination
Procedure: Conventional Venepuncture — This involves the conventional method of identifying veins suitable for venepuncture, which involves visualization and palpation.
  Arms: Conventional Venepuncture

SUMMARY:
Our novel technique of pen-torch transillumination (PTI) uses a cheap and easily available instrument (Penlite-LP212®, Energizer®, Missouri, USA) to visualize superficial veins invisible to the naked eye. The investigators evaluate the efficacy of PTI in improving venepuncture success rate (SR) for patients with poor venous access.

This prospective randomized controlled trial looks at adult patients aged 21 to 90 with difficult venous access (history of ≥3 consecutive attempts required for successful cannulation during the current admission) requiring non-emergent venepuncture. Patients will undergo venepuncture over the upper-limb using one of the following: Conventional venepuncture (control); Veinlite® (TransLite®, Texas, USA), a commercial transillumination device; PTI. Outcome measures are: successful cannulation within 2 attempts; duration of each successful attempt. Fisher's exact and Kruskal-Wallis tests will be performed.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial. Patients with a history of difficult venepuncture who agree to be entered into the study will be randomized into one of 3 groups using a sealed envelope system: 1. Conventional venepuncture (Control Group, n=25); 2. Veinlite® a commercial LED transilluminator device (Experimental Group 1, n=25); 3. Pen torch transillumination (Experimental Group 2, n=25). Hemodynamically unstable patients are excluded. The nurse involved in the care of the patient will attempt venepuncture over the upper limb. A maximum of 4 times attempts is allowed, before escalation to a doctor/phlebotomist.

A standardized venepuncture technique using standardized instruments will be utilized. Veins will be localized using one of the above techniques. Pen torch transillumination and veinlite are non-invasive techniques for locating veins. For pen torch transillumination, the tip of the pen torch is pressed onto the skin, causing the shadow of the vein to show up. Veinlite uses a device that emits red light. Placing it onto the skin will cause the outlines of the veins to show up. Once a suitable vein is localized, a tourniquet is applied (Braun® International, USA). The area of the skin to be cannulated is disinfected with an alcohol wipe (Webcol®, Covidien®, USA). For the setting of IV cannulation, a standardized 23G IV cannula is used (Introcan Safety®, Braun®, USA). Normal saline (PosiFlush® 3ml, BD®, USA) will be used for flushing the cannula after successful cannulation. For blood taking, a syringe (Terumo®, Philippines) ranging from 2ml to 20ml and a 23G needle (Venofix®, Braun®, USA) will be used. All instruments needed for venepuncture, including 4 IV cannula or 4 needles should be by the patient's bedside prior to the start of each venepuncture.

Duration of the procedure will be recorded using a stop watch. This is defined as the time (in minutes) from the start of attempt to localize a vein to its successful cannulation. Successful cannulation is defined either as the ability to flush 2ml of normal saline into the IV cannula or the ability to draw 2ml of blood from the vein.

A post-procedure questionnaire will be filled up by the nurses after attempt at venepuncture (refer to attached file). Outcome data include: number of attempts and duration needed for successful venepuncture. Patient data include: age, sex, race, body-mass index, history of intra-venous drug abuse, and renal function.

ELIGIBILITY:
Inclusion Criteria:

* History of ≥3 consecutive attempts required for successful cannulation during the current admission
* Patients requiring non-emergent venous cannulation for blood sampling or intra-venous plug insertion

Exclusion Criteria:

* Patients who are haemodynamically unstable

Respiratory Rate (< 8 or > 30 / min) SpO2 (< 93% on max 4L O2 on NP) Pulse rate (< 40 or > 130 bpm) Blood pressure (SBP < 90 mmHg) Acute change in mental state

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of venepuncture attempts | 1 day
  We record the number of attempts required for successful venepuncture

SECONDARY OUTCOMES:
Duration of venepuncture | 1 day
  A stopwatch will be used to measure the duration required from the start of vein identification, to the end of a successful venepuncture attempt.

CONTACTS AND LOCATIONS:
Overall Officials: Thiam Chye Lim, FRCS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Result] Katsogridakis YL, Seshadri R, Sullivan C, Waltzman ML. Veinlite transillumination in the pediatric emergency department: a therapeutic interventional trial. Pediatr Emerg Care. 2008 Feb;24(2):83-8. doi: 10.1097/PEC.0b013e318163db5f. PMID 18277843
- [Result] Yen K, Gorelick MH. New biomedical devices that use near-infrared technology to assist with phlebotomy and vascular access. Pediatr Emerg Care. 2013 Mar;29(3):383-5; quiz 386-7. doi: 10.1097/PEC.0b013e31828680f9. PMID 23462399
- [Result] Mbamalu D, Banerjee A. Methods of obtaining peripheral venous access in difficult situations. Postgrad Med J. 1999 Aug;75(886):459-62. doi: 10.1136/pgmj.75.886.459. PMID 10646021